CLINICAL TRIAL: NCT00185042
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study of the Efficacy and Safety of the ACAT Inhibitor CS-505 for Reducing the Progression of Atherosclerosis in Subjects With Coronary Artery Disease Using Intravascular Ultrasound (IVUS)
Brief Title: Efficacy and Safety of the ACAT Inhibitor CS-505 (Pactimibe) for Reducing the Progression of Coronary Artery Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 505-202
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Last update posted 2007-09-11 (Estimated); Status verified 2007-09

CONDITIONS: Coronary Heart Disease
Keywords: Atherosclerosis, intravascular ultrasound
MeSH Terms: conditions — Coronary Disease; Atherosclerosis | interventions — pactimibe

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

INTERVENTIONS:
Drug: Pactimibe, CS-505

SUMMARY:
The purpose of this study is to learn if CS-505 is safe and effective for slowing down or possibly reversing the buildup of tissue, cells and fatty deposits (plaque) in the blood vessels of the heart (coronary artery atherosclerosis).

ELIGIBILITY:
Inclusion Criteria:

Standard:

1. Male or female subjects, age 18 years or greater; and
2. Diagnosed or suspected coronary artery disease with a clinical indication for coronary angiography.

Angiographic:

1. Evidence of coronary heart disease
2. Identification of a target native coronary artery for the plaque volume measurement.

Exclusion Criteria:

Standard:

1. Breast feeding or lactating women, or women who have had a pregnancy (regardless of outcome) within the past 12 months;
2. Previous heart or other organ transplantation;
3. Treatment with any of the following agents within 4 weeks prior to randomization:

   * Immunosuppressive agents (cyclosporine, azathioprine);
   * Rifampin; and
   * Phenytoin, phenobarbital, valproic acid, or other anticonvulsants.
4. Any of the following manifestations of cardiac disease:

   * Myocardial infarction or unstable angina within 24 hours prior to randomization or clinically unstable;
   * Clinically significant heart disease; and
   * Coronary artery bypass surgery within previous 3 months.
5. Stroke (CVA) within previous 3 months;
6. Evidence of severe symptomatic heart failure (NYHA Class III or IV) or known ejection fraction less than 30%;
7. Uncontrolled diabetes mellitus;
8. Uncontrolled hypertension; and
9. Nephrotic syndrome, significant nephropathy, or other significant renal disease.

Angiographic:

1. Presence of any lesion with greater than 50% reduction in lumen diameter; or
2. Any lesion with a greater than 50% occlusion in the left main coronary artery;
3. A target vessel, including any of its branches, that has undergone or will be undergoing coronary artery bypass grafting (CABG) or percutaneous coronary intervention (PCI);
4. A target vessel that is itself a bypass graft.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 534 (Actual)
Dates: Start 2002-11; Study Completion 2005-07

PRIMARY OUTCOMES:
To compare the effect of CS-505 versus placebo when added to usual medical care on the change from baseline in percent atheroma volume, as measured by intravascular ultrasound (IVUS) of the identified target coronary artery segment

SECONDARY OUTCOMES:
To compare the effect of CS-505 versus placebo when added to usual medical care on:
- change from baseline in total atheroma volume in
various arteries;
- changes in minimum luminal diameter and percent
diameter stenosis;
- incidence and time to first occurrence of
cardiovascular events.
To compare the safety of CS-505 versus placebo

CONTACTS AND LOCATIONS:
Locations (46):
- United States (46):
  - Birmingham, Alabama
  - Huntsville, Alabama
  - Mobile, Alabama
  - Phoenix, Arizona
  - Los Angeles, California
  - San Diego, California
  - Fort Collins, Colorado
  - Bridgeport, Connecticut
  - Newark, Delaware
  - Clearwater, Florida
  - Gainsville, Florida
  - Hudson, Florida
  - Jacksonville, Florida
  - Melbourne, Florida
  - Miami, Florida
  - Pensacola, Florida
  - Port Charlotte, Florida
  - Sarasota, Florida
  - Tallahassee, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Springfield, Illinois
  - Louisville, Kentucky
  - Baltimore, Maryland
  - Springfield, Massachusetts
  - Grand Rapids, Michigan
  - Kalamazoo, Michigan
  - Duluth, Minnesota
  - Minneapolis, Minnesota
  - Kansas City, Missouri
  - Lincoln, Nebraska
  - New York, New York
  - Rochester, New York
  - Troy, New York
  - Charlotte, North Carolina
  - Greenville, North Carolina
  - High Point, North Carolina
  - Winston-Salem, North Carolina
  - Akron, Ohio
  - Cleveland, Ohio
  - Elyria, Ohio
  - Mansfield, Ohio
  - Oklahoma City, Oklahoma
  - Doylestown, Pennsylvania
  - Memphis, Tennessee
  - San Antonio, Texas

REFERENCES:
- [Derived] Nissen SE, Tuzcu EM, Brewer HB, Sipahi I, Nicholls SJ, Ganz P, Schoenhagen P, Waters DD, Pepine CJ, Crowe TD, Davidson MH, Deanfield JE, Wisniewski LM, Hanyok JJ, Kassalow LM; ACAT Intravascular Atherosclerosis Treatment Evaluation (ACTIVATE) Investigators. Effect of ACAT inhibition on the progression of coronary atherosclerosis. N Engl J Med. 2006 Mar 23;354(12):1253-63. doi: 10.1056/NEJMoa054699. PMID 16554527